CLINICAL TRIAL: NCT06679101
Title: A Phase 3, Randomized, Open-label Study of Belantamab Mafodotin Administered in Combination With Lenalidomide and Dexamethasone (BRd) Versus Daratumumab, Lenalidomide, and Dexamethasone (DRd) in Participants With Newly Diagnosed Multiple Myeloma Who Are Ineligible for Autologous Stem Cell Transplantation (TI-NDMM)
Brief Title: A Study of Belantamab Mafodotin Administered in Combination With Lenalidomide and Dexamethasone (BRd) Versus Daratumumab, Lenalidomide, and Dexamethasone (DRd) in Participants With Newly Diagnosed Multiple Myeloma (NDMM) Who Are Ineligible for Autologous Stem Cell Transplantation (TI-NDMM)
Acronym: DREAMM-10
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 214828; 2024-516030-35 (Registry Identifier: CTIS)
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma; Newly Diagnosed Multiple Myeloma
Keywords: Multiple myeloma; Belantamab mafodotin; Lenalidomide; Dexamethasone; Daratumumab; Transplant-ineligible; DREAMM-10
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin; Lenalidomide; Dexamethasone; daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Belantamab Mafodotin + Lenalidomide + Dexamethasone (Experimental): Belantamab mafodotin, lenalidomide, and dexamethasone will be administered.
  Treatment will continue in both arms until progressive disease (PD), death, unacceptable toxicity, withdrawal of consent, or end of study, whichever occurs first.
  Interventions: Drug: Belantamab mafodotin; Drug: Lenalidomide; Drug: Dexamethasone
- Arm B: Daratumumab + Lenalidomide + Dexamethasone (Active Comparator): Daratumumab, lenalidomide, and dexamethasone will be administered.
  Treatment will continue in both arms until PD, death, unacceptable toxicity, withdrawal of consent, or end of study, whichever occurs first.
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone; Drug: Daratumumab

INTERVENTIONS:
Drug: Belantamab mafodotin — Belantamab mafodotin will be administered.
  Arms: Arm A: Belantamab Mafodotin + Lenalidomide + Dexamethasone
Drug: Lenalidomide — Lenalidomide will be administered.
Drug: Dexamethasone — Dexamethasone will be administered.
Drug: Daratumumab — Daratumumab will be administered.
  Arms: Arm B: Daratumumab + Lenalidomide + Dexamethasone

SUMMARY:
The purpose of this Phase 3 study is to evaluate if BRd prolongs progression free survival (PFS) and/or improves minimal residual disease (MRD) negative status compared with DRd in participants with TI-NDMM.

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 18 or the legal age of consent in the jurisdiction in which the study is taking place, at the time of signing the informed consent.
2. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form and in the protocol.
3. NDMM with a requirement for treatment as documented per IMWG criteria.
4. Must have at least 1 aspect of measurable disease, as assessed by the central laboratory, defined as 1 of the following:

   1. Urine M-protein excretion ≥200 mg/24 hours (≥0.2 g/24 hours) And/or
   2. Serum M-protein concentration ≥0.5 g/dL (≥5.0 g/L) And/or
   3. Serum free light-chain (FLC) assay: involved FLC level ≥10 mg/dL (≥100 mg/L) and an abnormal serum FLC ratio (<0.26 or >1.65).
5. Newly diagnosed and not considered candidate for high-dose chemotherapy with autologous stem cell transplant (ASCT) due to any of the following:

   1. ≥70 years of age, OR
   2. Age 18 to 69 years with presence of comorbid condition(s) likely to have a negative impact on tolerability of high-dose chemotherapy with ASCT, (or for whom national guidelines do not permit transplant due to a cut-off age below 70 years), OR
   3. Who refuse high-dose chemotherapy with ASCT as an initial treatment.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
7. Adequate organ system function as defined by the laboratory assessments.
8. Male participants:

   * Contraceptive use by men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
   * Male participants are eligible to participate if they agree to the following during the Treatment Period and for at least 6 months after the last dose of study intervention to allow for clearance of any altered sperm:
   * Refrain from donating fresh unwashed semen

   PLUS either:
   * Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent.

   OR
   * Must agree to use contraception/barrier as detailed below
   * Agree to use a male condom, even if they have undergone a successful vasectomy, and female partner to use an additional highly effective contraceptive method with a failure rate of <1% per year when having sexual intercourse with a woman of childbearing potential (WOCBP) who is not currently pregnant. Male participants should also use a condom when having sexual intercourse with pregnant females.
9. Female participants

   * Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
   * A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least 1 of the following conditions applies:
   * Is not a WOCBP OR
   * Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), preferably with low user dependency during the Treatment Period and for 4 months after the last dose of study intervention and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention.
   * A WOCBP must have 2 negative highly sensitive serum pregnancy tests before starting treatment, the first may be performed within 14 days from C1D1, the second within 24 hours before the first dose of study intervention.
   * Should pregnancy occur in a female on treatment or the female partner of a male on treatment, treatment must be stopped, and it is advised to seek advice from a physician specialized or experienced in teratology.

Exclusion Criteria:

1. Diagnosis of systemic amyloid light chain amyloidosis, Waldenstrom's disease, POEMS (polyneuropathy, organomegaly, endocrinopathy, monoclonal plasma proliferative disorder, skin changes) or Primary Plasma Cell Leukemia (defined as circulating plasma cells >5%).
2. Prior systemic therapy for multiple myeloma, or smoldering multiple myeloma.
3. Signs of meningeal or central nervous system involvement with multiple myeloma.
4. Major surgery within 2 weeks prior to the first dose of study drugs or has not recovered fully from surgery. Kyphoplasty is not considered major surgery.
5. Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions (including lab abnormalities) that could interfere with participant's safety, obtaining informed consent, or compliance with study procedures.
6. Current active liver or biliary disease (except for Gilbert's syndrome or asymptomatic gallstones, or otherwise stable chronic liver disease as per the investigator's assessment).
7. Participants with previous or concurrent malignancies other than multiple myeloma are excluded. Exceptions are any other malignancy that has been considered medically stable for at least 2 years, after discussion with the GSK Medical Monitor. The participant must not be receiving active therapy, other than hormonal therapy for this disease.
8. Evidence of cardiovascular risk including any of the following:

   1. Evidence of current clinically significant untreated arrhythmias, including clinically significant electrocardiogram abnormalities including second-degree (Mobitz Type II) or third-degree atrioventricular block.
   2. Recent history (within 3 months of screening) of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty or stenting, or bypass grafting.
   3. Class III or IV heart failure as defined by the New York Heart Association functional classification system.
9. Known human immunodeficiency virus (HIV) infection, unless the participant can meet all of the following criteria:

   1. Established antiretroviral therapy for at least 4 weeks and HIV viral load <400 copies/mL within Screening Period.
   2. CD4+ T-cell (CD4+) counts ≥350 cells/μL.
   3. No history of acquired immune deficiency syndrome-defining opportunistic infections within the last 12 months.
10. Positive hepatitis C antibody test result or positive hepatitis C ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study intervention unless the participant can meet the following criteria:

    1. RNA test negative.
    2. Successful antiviral treatment (usually 8 weeks duration) is required, followed by a negative hepatitis C viral load RNA test after a washout period of at least 4 weeks.
11. Participants with hepatitis B will be excluded unless the defined criteria can be met.
12. Current corneal epithelial disease except for mild punctate keratopathy.
13. Intolerance or contraindications to antiviral prophylaxis.
14. Unable to tolerate antithrombotic prophylaxis.
15. Known immediate or delayed hypersensitivity reaction or idiosyncratic reaction to drugs chemically related to belantamab mafodotin, or any of the components of the study intervention.
16. Plasmapheresis within 7 days prior to the first dose of study intervention.
17. Participants must not have received a live or live-attenuated vaccine within 30 days prior to first dose of belantamab mafodotin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2031-03-31 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
PFS | Up to approximately 7 years
  Defined as the time from the date of randomization to the date of first documented PD per International Myeloma Working Group (IMWG) criteria by Independent Review Committee (IRC) or death from any cause in the absence of progression, whichever occurs first.
Number of Participants Achieving MRD Negative Status | Up to approximately 7 years
  Defined as achieving MRD negativity at 10^-5 sensitivity threshold (1 nucleated tumor cell in 100,000 normal cells) assessed by next-generation sequencing (NGS) at least once during the time of confirmed complete response (CR) or better response per IMWG criteria by IRC.

SECONDARY OUTCOMES:
PFS2 | Up to approximately 7 years
  Defined as the time from the date of randomization to the date of documented PD following the first subsequent anti-myeloma therapy or death from any cause, whichever is earlier.
Overall Survival (OS) | Up to approximately 7 years
Number of Participants Achieving CR or Better (CR+) | Up to approximately 7 years
Number of Participants Achieving Very Good Partial Response (VGPR) or Better | Up to approximately 7 years
Number of Participants Achieving Sustained MRD Negative Status | Up to approximately 7 years
  Defined as achieving MRD negative status at 10^-5 sensitivity threshold (1 nucleated tumor cell in 100,000 normal cells) assessed by NGS at least twice, a minimum of 1 year apart and with no MRD positive result in between, during the time of confirmed CR+ response per IMWG criteria by IRC.
Duration of Response (DoR) | Up to approximately 7 years
Time to Second Next Line Therapy (TTST) | Up to approximately 7 years
Number of Participants With Adverse Events (AEs) | Up to approximately 7 years
Number of Participants With Ocular Findings on Ophthalmic Exam | Up to approximately 7 years
Maximum Post-baseline Patient-Reported Outcomes Version of the Common Term Criteria for Adverse Events (PRO-CTCAE) Score | Up to approximately 7 years
Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ)-C30 | Up to approximately 7 years
Change From Baseline in EORTC QLQ-MY20 | Up to approximately 7 years
Plasma Concentrations of Belantamab Mafodotin | Up to approximately 7 years
Number of Participants With Positive Anti-drug Antibodies (ADAs) Against Belantamab Mafodotin | Up to approximately 7 years
Titers of ADAs Against Belantamab Mafodotin | Up to approximately 7 years

CONTACTS AND LOCATIONS:
Locations (156):
- United States (24):
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Pasadena, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Englewood, Florida
  - GSK Investigational Site, Lady Lake, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Saint Augustine, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Portland, Maine
  - GSK Investigational Site, Worcester, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Billings, Montana
  - GSK Investigational Site, Stony Brook, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Kingwood, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, Fairfax, Virginia
- Argentina (5):
  - GSK Investigational Site, Capital Federal
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aire
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Rosario
  - GSK Investigational Site, Viedma
- Australia (6):
  - GSK Investigational Site, Gosford NSW, New South Wales
  - GSK Investigational Site, Box Hill, Victoria
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Fitzroy
  - GSK Investigational Site, Herston
  - GSK Investigational Site, St Leonards
- Belgium (5):
  - GSK Investigational Site, Bruges
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Hornu
  - GSK Investigational Site, Roeselare
- Brazil (8):
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Barretos
  - GSK Investigational Site, Joinville
  - GSK Investigational Site, Porto Alegre
  - GSK Investigational Site, Salvador
  - GSK Investigational Site, São Paulo
  - GSK Investigational Site, Teresina
  - GSK Investigational Site, Vitória
- GSK Investigational Site, Saint John, New Brunswick, Canada
- China (12):
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Chengdu
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Nanchang
  - GSK Investigational Site, Nanjing
  - GSK Investigational Site, Shanghia
  - GSK Investigational Site, Shenzhen
  - GSK Investigational Site, Tianjin
  - GSK Investigational Site, Wenzhou
  - GSK Investigational Site, Xi'an
- Czechia (2):
  - GSK Investigational Site, Ostrava
  - GSK Investigational Site, Prague
- France (3):
  - GSK Investigational Site, Bobigny
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Villejuif
- Germany (9):
  - GSK Investigational Site, Jena, Europe
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Chemnitz
  - GSK Investigational Site, Cologne
  - GSK Investigational Site, Dresden
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Hanover
  - GSK Investigational Site, Mainz
  - GSK Investigational Site, Würzburg
- Greece (4):
  - GSK Investigational Site, Alexandroupoli
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Pátrai
  - GSK Investigational Site, Thessaloniki
- India (6):
  - GSK Investigational Site, Ahmedabad
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Hyderabad
  - GSK Investigational Site, Kolkata
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Sushrut Hospital and Research
- Ireland (3):
  - GSK Investigational Site, Dublin
  - GSK Investigational Site, Galway
  - GSK Investigational Site, Waterford
- Israel (5):
  - GSK Investigational Site, Beersheba
  - GSK Investigational Site, Jerusalem
  - GSK Investigational Site, Koranit
  - GSK Investigational Site, Petah Tikva
  - GSK Investigational Site, Tel Aviv
- Italy (7):
  - GSK Investigational Site, Ancona
  - GSK Investigational Site, Catania
  - GSK Investigational Site, Meldola FC
  - GSK Investigational Site, Palermo
  - GSK Investigational Site, Pavia
  - GSK Investigational Site, Pisa
  - GSK Investigational Site, Roma
- Japan (18):
  - GSK Investigational Site, Shibuya-Ku, Tokyo
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Fukushima
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Ishikawa
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Nara
  - GSK Investigational Site, Numakunai
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Sapporo
  - GSK Investigational Site, Suita
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Yamagata
- Norway (3):
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Lrenskog
  - GSK Investigational Site, Oslo
- Poland (4):
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wałbrzych
- South Africa (2):
  - GSK Investigational Site, Kuils River
  - GSK Investigational Site, Pretoria
- South Korea (4):
  - GSK Investigational Site, Hwasun
  - GSK Investigational Site, Jeonju
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Ulsan
- Spain (9):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Gijón
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Salamanca
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Valladolid
- Taiwan (5):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Tainan
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan District
- Turkey (Türkiye) (6):
  - GSK Investigational Site, Samsun, Atakum
  - GSK Investigational Site, Kocaeli, İzmit
  - GSK Investigational Site, Ankara, Yenimahalle
  - GSK Investigational Site, Adana
  - GSK Investigational Site, Ankara
  - GSK Investigational Site, Sisli - Istanbul
- United Kingdom (5):
  - GSK Investigational Site, Leicester
  - GSK Investigational Site, Middlesbrough
  - GSK Investigational Site, Oxford
  - GSK Investigational Site, Plymouth
  - GSK Investigational Site, Wolverhampton

IPD SHARING:
Plan to Share IPD: No
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.